CLINICAL TRIAL: NCT01956565
Title: Feasibility of Inspiratory Muscle Training in People With Chronic Obstructive Pulmonary Disease (COPD) Who Decline Pulmonary Rehabilitation
Brief Title: Feasibility of Inspiratory Muscle Training in People With COPD Who Decline Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STH 16453
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Rehabilitation; Physiotherapy; Patient Compliance; Inspiratory Muscle Training; Respiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory muscle training (Experimental): Participants will perform 8 weeks of IMT strength training using the Powerbreathe Kinetic device (Powerbreathe). Training will progress to 60% maximum inspiratory pressure (PiMax) with 30 breaths at high velocity (paced initially over a period of 15 minutes), twice a day, 5 days per week. Tidal breathing without inspiratory resistance is acceptable for recovery between each high velocity breath. Training will be titrated and supervised weekly for the first 8 weeks by a physiotherapist. After 8 weeks training the participants are advised to continue training unsupervised, twice a day, 3 times per week for a further 18 weeks.
  Interventions: Other: Inspiratory Muscle training
- Declining Inspiratory muscle training (No Intervention): No intervention. Interview and baseline assessment only.

INTERVENTIONS:
Other: Inspiratory Muscle training — Participants will perform 8 weeks of IMT strength training using the Powerbreathe Kinetic device (Powerbreathe). Training will progress to 60% maximum inspiratory pressure (PiMax) with 30 breaths at high velocity (paced initially over a period of 15 minutes), twice a day, 5 days per week. Tidal breathing without inspiratory resistance is acceptable for recovery between each high velocity breath. Training will be titrated and supervised weekly for the first 8 weeks by a physiotherapist. After 8 weeks training the participants are advised to continue training unsupervised, twice a day, 3 times per week for a further 18 weeks.
  Arms: Inspiratory muscle training

SUMMARY:
The feasibility study will involve mixed methods, this means interviews as well as assessment of treatment with inspiratory muscle training therapy (IMT). There are two pathways within the study depending on whether people want to have inspiratory muscle training. People who accept to have inspiratory muscle training will have assessments before training, after 8 weeks of training and at 6 month follow up in addition to interviews before and after the study (at 6 months). For those who choose not to have the inspiratory muscle training the investigators will offer them an interview so that the investigators can find out more about what might have made the study more appealing or what treatments they would have preferred. The investigators will also ask if they wish to be followed up with baseline assessments for the study period and if the investigators can access health records.

Interviews

Semi-structured interviews lasting approximately an hour will be performed at the beginning of the study with participants who accept the IMT pathway and those who decline IMT until no knew themes are raised. These interviews will be used to provide information on reasons for declining pulmonary rehabilitation, attitudes to exercise, attitudes to IMT, treatment preferences and opinions regarding study design and outcome measures (see Interview Topic guide). The interviews will be taped and transcribed verbatim. A follow up interview with study participants who have received IMT will be conducted at 6 months addressing attitudes to IMT and study design and whether they have decided that they wish to engage with other services (such as pulmonary rehabilitation and smoking cessation).

Inspiratory Muscle Training (IMT) method

Participants will perform 8 weeks of IMT strength training using the Powerbreathe Kinetic device (Powerbreathe). Training will progress to 60% maximum inspiratory pressure (PiMax). This means that each breath in through the device is set at 60% of the maximum force you are able to create when you breathe in rather than at full force. 30 breaths are performed at high velocity (paced initially over a period of 15 minutes to allow recovery between each breath through the device). Once established it is anticipated that each training session should take no more than five minutes. Training is performed twice a day, 5 days per week for the first 8 weeks. Training will be titrated (set to a level suitable for the participant) and supervised weekly for the first 8 weeks by a physiotherapist. After 8 weeks training the participants are advised to continue training unsupervised, twice a day, 3 times per week for a further 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 35
* with stable COPD (having had no exacerbation needing antibiotics or steroids in the preceding four weeks) with breathlessness on Medical Research Council (MRC) scale of 3 or above who decline Pulmonary rehabilitation (MRC 3 is defined as "walks slower than contemporaries on level ground because of breathlessness, or has to stop for breath when walking at own pace").

Exclusion Criteria:

* History of spontaneous pneumothorax
* incomplete recovery from a traumatic pneumothorax
* asthma
* known recently perforated eardrum
* unstable angina
* ventricular dysrhythmias
* cerebral event or myocardial infarction within the last two months
* not oral antibiotics or steroids for COPD exacerbation within the last four weeks

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recruitment | 4 months
  Recruitment of 10 participants for inspiratory muscle training and 10 participants for interview alone within a four month period.

SECONDARY OUTCOMES:
Adherence with Inspiratory muscle training | 6 months
  Adherence to IMT: measured using a customised electronic threshold device (Powerbreathe) recording data from baseline to 6 months. Adherence will also be assessed using participant diaries.
Attrition rate. | 6 months
  Attrition rate over the 6 month course of treatment.
Maximal inspiratory pressure (PiMax) | Baseline, 8 weeks, 6 months
  Inspiratory muscle strength: Maximal inspiratory pressure (PiMax) and Sniff Nasal pressure measured using the MicroRPM (Micromedical) at baseline, 8 weeks and 6 months.
Acceptability | 6 months
  Acceptability of IMT, study design and outcome measures and engagement or intention to engage with other services will be addressed in interviews at baseline and at 6 months for participants. A single interview will be offered to those declining the IMT arm of the study.

OTHER OUTCOMES:
Health related quality of life (HRQOL) | Baseline, 8 weeks, 6 months
  HRQOL measured using the Chronic Respiratory Disease questionnaire (CRQ) and COPD Assessment Test.
Anxiety and depression | Baseline, 8 weeks, 6 months
  Anxiety and depression measured using the Hospital Anxiety and Depression Questionnaire.
Activity Monitory | Baseline, 8 weeks, 6 months
  Activity monitoring assessed using Sensewear Accelerometers (Sensewear Pro-Armband Bodymedia) worn for four days.
Dyspnoea | Baseline, 8 weeks, 6 months
  Dyspnoea measured using the first 5 questions of the CRQ. Dyspnoea will also be measured by the modified BORG breathlessness score recorded pre and post IMT.
Healthcare utilisation | 6 months
  Healthcare utilisation measured using patient diaries and electronic health records, and EQ5DL.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Services, Sheffield Teaching Hospitals, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] O'Connor C, Lawson R, Waterhouse J, Mills GH. Is inspiratory muscle training (IMT) an acceptable treatment option for people with chronic obstructive pulmonary disease (COPD) who have declined pulmonary rehabilitation (PR) and can IMT enhance PR uptake? A single-group prepost feasibility study in a home-based setting. BMJ Open. 2019 Aug 8;9(8):e028507. doi: 10.1136/bmjopen-2018-028507. PMID 31399454